CLINICAL TRIAL: NCT02141555
Title: Comparing Buccal and Vaginal Misoprostol in Management of Early Pregnancy Loss: a Pilot Randomized Controlled Trial
Brief Title: Comparing Buccal and Vaginal Misoprostol in Management of Early Pregnancy Loss
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheila Mody, Assistant Adjunct Professor, Section of Family Planning, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140250
Record Dates: First submitted 2014-05-10; First posted 2014-05-19 (Estimated); Results first posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-07

CONDITIONS: Spontaneous Abortion in First Trimester
Keywords: misoprostol, early pregnancy loss, missed abortion
MeSH Terms: conditions — Abortion, Spontaneous; Abortion, Missed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaginal misoprostol (Active Comparator): Participants will insert four misoprostol tablets (total of 800 micrograms) deeply into the vagina with their fingers.
  Interventions: Drug: Vaginal Misoprostol
- Buccal Misoprostol (Experimental): Participants will place two tablets of misoprostol between their gum and cheek on each side (total 800 micrograms), then swish and swallow the remnants after 30 minutes.
  Interventions: Drug: Buccal Misoprostol

INTERVENTIONS:
Drug: Vaginal Misoprostol — Misoprostol inserted into vagina
  Other Names: Vaginal Cytotec
  Arms: Vaginal misoprostol
Drug: Buccal Misoprostol — Misoprostol placed between the gum and cheek and allowed to dissolve for 30 minutes with the remnants swallowed after this time.
  Other Names: Buccal Cytotec
  Arms: Buccal Misoprostol

SUMMARY:
First trimester miscarriages are common. When the failed pregnancy does not pass spontaneously on its own, it is called a missed abortion. There are several ways in which missed abortions are managed, one of which involves administering a medication called misoprostol which causes uterine contractions inducing expulsion of the failed pregnancy. Misoprostol can be administered in multiple ways but has been traditionally inserted vaginally when used for management of missed abortions. Some studies have shown that some women are not comfortable with vaginal insertion of misoprostol and prefer oral administration. Buccal misoprostol is a way of administering misoprostol by having the patients insert the tablets of misoprostol between their gum and cheek, letting it dissolve for 30 minutes, then swallowing the remaining remnants. Buccal misoprostol is used safely in medical abortion. In fact a study by Fjerstad et al (2009), found a decrease in infection rate for medical abortion when misoprostol administration was switched from vaginal to buccal route combined with routine administration of doxycycline. The efficacy of using buccal misoprostol to treat missed abortions has not been studied previously to the investigators' knowledge. In this pilot study, investigators aim to test the hypotheses that buccal misoprostol is equally effective as vaginal misoprostol in the medical management of early pregnancy loss. As secondary outcomes, investigators suspect that buccal misoprostol may be associated with higher rates of gastrointestinal side effect but that patient satisfaction will remain equally as high for buccal misoprostol as for vaginal misoprostol.

DETAILED DESCRIPTION:
Randomization:

Women who present to University of California, San Diego (UCSD) Medical Offices South clinic for evaluation and management of missed abortion will all be sent to the lab prior to the clinic visit for a type and screen and hemogram to determine blood type and hemoglobin level as is the current standard of care. Each woman will then be screened by a physician. The physician will notify a co-investigator of eligible patients who are interested in participating in the study. The co-investigator will consent the patient for the study. Once the written consent is obtained, patient will be asked to fill out an intake survey to obtain demographic information. Participants will be randomized into either the vaginal or buccal misoprostol group with a block size of four. Assignments will be concealed in sequentially numbered sealed opaque envelope. The envelope will be opened by the co-investigator who will reveal the route of misoprostol to the patient and review the written instructions on how to take the medication appropriately. Given the different routes of administration, neither the patient nor the provider will be blinded. Given that one of the secondary outcomes of interest was patient satisfaction based on the different route of administration, decision was made to not use placebo pills which could have been used to do a double-blinded study.

Intervention:

Dose of Misoprostol for both treatment groups: 800 micrograms administered as four tablets of 200 micrograms.

Currently, the standard of care is to prescribe vaginal misoprostol 800 mcg for women with an early pregnancy failure desiring medical management. The only "intervention" in this study is to change the route of administration from vaginal to buccal for the women randomized to this group. The dose of misoprostol, follow up plan (including ultrasound) and prescription for pain medications (described below) is unchanged from the current standard of care. Participants randomized to the vaginal misoprostol group will be instructed to insert four misoprostol tablets (total of 800 micrograms) deeply into the vagina with their fingers. Participants randomized to the buccal misoprostol group will be instructed to place two tablets of misoprostol between their gum and cheek on each side (total 800 micrograms), then swish and swallow the remnants after 30 minutes. If the patient is Rh negative, the patient will be given a dose of rhogam 300 mcg at the initial visit which is the current standard of care.

Patients will be prescribed an additional dose of misoprostol 800 mcg that they can take at their own discretion in the absence of vaginal bleeding 48 hours from initial dose using the same route of administration as the first dose. All participants will be prescribed ibuprofen with instructions to take 600 mg every 6 hours as needed for pain and a narcotic medication for breakthrough pain. The cost of these medications will be fully covered by the participant's insurance with no additional cost to the participant.

Follow up will be a clinic visit scheduled one week from the from the initial visit at UCSD Medical Offices South Clinic which time the participant will fill out a follow up survey assessing the participant's satisfaction and side effects experienced. The provider will also fill out a survey at this 1-week follow up visit assessing the success of the misoprostol in achieving a complete abortion. The participant's involvement in the study will conclude at this end of this one-week follow up visit.

Participant Commitment:

The research will require the following additional time commitment from participant in addition to the standard clinic visit:

1. Initial Visit: An additional 20 minutes will be required to review the study consent, randomize to the vaginal or buccal misoprostol group, and have the patient fill out a short intake survey.
2. Follow-up visit: The follow up visit will take one week from time of initial visit. An additional 10 minutes will be required to fill out the follow up survey. The participant's involvement in the study will conclude with this visit.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 18-50 who are English or Spanish speaking
* First trimester pregnancy (less than 13 weeks and 0 days)
* Desires medical management of an early pregnancy loss with misoprostol
* Diagnosed with an early pregnancy failure by UCSD Radiology or diagnosed early pregnancy failure defined by any of the following criteria (Bourne 2013):

  * Crown-rump length > 7mm with no cardiac activity
  * Mean gestational sac diameter of > 25 mm and no embryo
  * Absence of an embryo with heartbeat > 2 weeks after a scan showing a gestational sac without a yolk sac
  * Absence of embryo with heartbeat > 11 days after a scan showing a gestational sac with a yolk sac

Exclusion Criteria:

* Evidence of infection, acute hemorrhage, or hemodynamic instability
* Hemoglobin less than 9.5 including use of point of care Hgb testing
* Known allergy to misoprostol
* Underwent surgical or medical abortion during current pregnancy
* Currently breastfeeding
* Currently has intrauterine device in place
* Suspicion of ectopic or gestational trophoblastic disease
* History of clotting disorder or on anticoagulant therapy (excluding aspirin)
* Unreliable for follow up

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janie Pak, MD, MPH, Study Director — University of California, San Diego; Sheila Mody, MD, MPH, Principal Investigator — University of California, San Diego
Locations (2):
- United States (2):
  - Universty of California San Diego Perlman Clinic, La Jolla, California
  - University of California San Diego Medical Offices South Clinic, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aronsson A, Fiala C, Stephansson O, Granath F, Watzer B, Schweer H, Gemzell-Danielsson K. Pharmacokinetic profiles up to 12 h after administration of vaginal, sublingual and slow-release oral misoprostol. Hum Reprod. 2007 Jul;22(7):1912-8. doi: 10.1093/humrep/dem098. Epub 2007 May 8. PMID 17488782
- [Background] Doubilet PM, Benson CB, Bourne T, Blaivas M; Society of Radiologists in Ultrasound Multispecialty Panel on Early First Trimester Diagnosis of Miscarriage and Exclusion of a Viable Intrauterine Pregnancy; Barnhart KT, Benacerraf BR, Brown DL, Filly RA, Fox JC, Goldstein SR, Kendall JL, Lyons EA, Porter MB, Pretorius DH, Timor-Tritsch IE. Diagnostic criteria for nonviable pregnancy early in the first trimester. N Engl J Med. 2013 Oct 10;369(15):1443-51. doi: 10.1056/NEJMra1302417. No abstract available. PMID 24106937
- [Background] Danielsson KG, Marions L, Rodriguez A, Spur BW, Wong PY, Bygdeman M. Comparison between oral and vaginal administration of misoprostol on uterine contractility. Obstet Gynecol. 1999 Feb;93(2):275-80. doi: 10.1016/s0029-7844(98)00436-0. PMID 9932569
- [Background] Fjerstad M, Trussell J, Sivin I, Lichtenberg ES, Cullins V. Rates of serious infection after changes in regimens for medical abortion. N Engl J Med. 2009 Jul 9;361(2):145-51. doi: 10.1056/NEJMoa0809146. PMID 19587339
- [Background] Jones RK, Kost K. Underreporting of induced and spontaneous abortion in the United States: an analysis of the 2002 National Survey of Family Growth. Stud Fam Plann. 2007 Sep;38(3):187-97. doi: 10.1111/j.1728-4465.2007.00130.x. PMID 17933292
- [Background] Herting RL, Clay GA. Overview of clinical safety with misoprostol. Dig Dis Sci. 1985 Nov;30(11 Suppl):185S-193S. doi: 10.1007/BF01309407. PMID 3932053
- [Background] Meckstroth KR, Whitaker AK, Bertisch S, Goldberg AB, Darney PD. Misoprostol administered by epithelial routes: Drug absorption and uterine response. Obstet Gynecol. 2006 Sep;108(3 Pt 1):582-90. doi: 10.1097/01.AOG.0000230398.32794.9d. PMID 16946218
- [Background] Middleton T, Schaff E, Fielding SL, Scahill M, Shannon C, Westheimer E, Wilkinson T, Winikoff B. Randomized trial of mifepristone and buccal or vaginal misoprostol for abortion through 56 days of last menstrual period. Contraception. 2005 Nov;72(5):328-32. doi: 10.1016/j.contraception.2005.05.017. Epub 2005 Aug 9. PMID 16246656
- [Background] Tang OS, Gemzell-Danielsson K, Ho PC. Misoprostol: pharmacokinetic profiles, effects on the uterus and side-effects. Int J Gynaecol Obstet. 2007 Dec;99 Suppl 2:S160-7. doi: 10.1016/j.ijgo.2007.09.004. Epub 2007 Oct 26. PMID 17963768
- [Background] Saraiya M, Berg CJ, Shulman H, Green CA, Atrash HK. Estimates of the annual number of clinically recognized pregnancies in the United States, 1981-1991. Am J Epidemiol. 1999 Jun 1;149(11):1025-9. doi: 10.1093/oxfordjournals.aje.a009747. PMID 10355378
- [Background] Schaff EA, DiCenzo R, Fielding SL. Comparison of misoprostol plasma concentrations following buccal and sublingual administration. Contraception. 2005 Jan;71(1):22-5. doi: 10.1016/j.contraception.2004.06.014. PMID 15639067
- [Background] Schaff EA, Fielding SL, Westhoff C. Randomized trial of oral versus vaginal misoprostol at one day after mifepristone for early medical abortion. Contraception. 2001 Aug;64(2):81-5. doi: 10.1016/s0010-7824(01)00229-3. PMID 11704083
- [Background] Sedgh G, Henshaw S, Singh S, Ahman E, Shah IH. Induced abortion: estimated rates and trends worldwide. Lancet. 2007 Oct 13;370(9595):1338-45. doi: 10.1016/S0140-6736(07)61575-X. PMID 17933648
- [Background] Wilcox AJ, Weinberg CR, O'Connor JF, Baird DD, Schlatterer JP, Canfield RE, Armstrong EG, Nisula BC. Incidence of early loss of pregnancy. N Engl J Med. 1988 Jul 28;319(4):189-94. doi: 10.1056/NEJM198807283190401. PMID 3393170
- [Background] Winikoff B, Dzuba IG, Creinin MD, Crowden WA, Goldberg AB, Gonzales J, Howe M, Moskowitz J, Prine L, Shannon CS. Two distinct oral routes of misoprostol in mifepristone medical abortion: a randomized controlled trial. Obstet Gynecol. 2008 Dec;112(6):1303-1310. doi: 10.1097/AOG.0b013e31818d8eb4. PMID 19037040

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 40 [31 to 49] | 35 [31 to 39] | 37.5 [31 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Patient Enrollment
Description: The percentage of women who are offered enrollment and accept.
Time Frame: One year
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

2. Secondary Outcome: Number of Participants With Complete Abortion
Description: Number of participants with complete abortion without surgical intervention defined as no evidence of a gestational sac on transvaginal ultrasound at the follow up visit.
Time Frame: one week
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol
Number analyzed (Participants) | 2 | 2
Participants | 1 | 2

3. Secondary Outcome: Number of Participants Who Answered 1 or 2 on a Scale of Satisfaction With the Procedure
Description: Written surveys patients will fill out at follow up visit assessing patient's satisfaction with the procedure.
  "How satisfied were you with your procedure?"
  The satisfaction scale used was:
  1 =Very Satisfied, comfortable, likely to recommend 3= Neutral 5= Very unsatisfied/uncomfortable, unlike to recommend
Time Frame: one week
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

4. Secondary Outcome: Number of Participants Reporting 2 or 3 on a Scale of Medication Side Effects
Description: Assessment of medication side effects including: nausea, vomiting, headache, fever (over 100.4 F), dizziness, diarrhea, bad taste, dry mouth "Did you experience any of these side effects? If so, how long did they last?"
  Patients asked on a scale of 0 to 3, where:
  Side Effect scale:
  0 = never
  1= less than one day 2 = 1 to 2 days 3 = more than 2 days
Time Frame: one week
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: One week
Arm/Group | Vaginal Misoprostol | Buccal Misoprostol
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Due to the small number of participants, no conclusions could be drawn and a larger study was not done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes